CLINICAL TRIAL: NCT02323308
Title: Study of Immunological, Virological, Serological Characteristics of HIV+ Patients Harboring Isolated Anti-HBc Profile and Response to Hepatitis B Vaccination
Brief Title: Isolated Anti-HBc Serological Profile in HIV Infected Patients: Immunological, Virological Characteristics and Response to Hepatitis B Vaccination
Acronym: ANRSHBEP03
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS HB EP 03 CISOVAC; 2010-A00511-38 (Other: ANSM)
Record Dates: First submitted 2014-07-11; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infection; Hepatitis B
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- vaccination: Anti-HBV vaccine injection
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling

SUMMARY:
The aim of study is to describe the clinical, immunological, serological, virological and therapeutic characteristics of HIV+ patients harboring isolated anti-HBc profile and to assess the response to vaccination in these patients.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ adults patients
* negative HBsAg
* negative a-HBs Ab
* positive HBc Ab
* without HBV - vaccination
* CD4 cell above 200 /mm3
* HIV viral load below 50 copies/mL

Exclusion Criteria:

* positive HBs antigenemia in the past
* transaminitis above fivefold upper normal limit
* PT<50% or Platelet <50 000/mm3
* ongoing opportunistic infection
* ongoing or recent systemic corticoid or immunomodulatory therapy, splenectomy, pregnancy, contra-indication to intramuscular injection, familial history of neurological disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with HIV infection and presenting with "isolated anti-HBc" profile. HBV vaccination is recommended fot these patients.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of immunological, virological and serological characteristics associated to "anti-HBc isolated" profile | at Day 0, inclusion visite
Average titers of anti-HBs Ab | at 4 weeks, 28 weeks and 18 months after the first vaccination HBV
Analysis of B-cell phenotype and maturation | at baseline and at week 28

SECONDARY OUTCOMES:
Number of patients with HBsAb titers as protective titer>10 IU/L | at 4 weeks,28 weeks and 18 month after the first dose HBV vaccin
Detection of IgG+ memory B cells specific for HBcAg or HBs Ag | at baseline and 28 weeks after the first dose HBV vaccin
- Detection of HBV preS2 and S-specific T cells | at day 0 and week 28

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Piroth, Principal Investigator — CHU DIJON
Locations (1):
- Chu Dijon, Dijon, France